CLINICAL TRIAL: NCT03137576
Title: Pain Blocks in Awake Thoracic Surgery: A Randomized Prospective Trial to Test the Non-inferiority of Erector Spinae Plane Block (ESPB) in Comparison With Paravertebral Block During Non-intubate, Thoracoscopic Lung Resection.
Brief Title: Erector Spinae Plane Block Versus Paravertebral Block During Non-intubated Thoracoscopic Lung Resections.
Acronym: PABATS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruiting and transfer of the PI to another center
Sponsor: IRCCS Sacro Cuore Don Calabria di Negrar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHT02
Record Dates: First submitted 2017-04-28; First posted 2017-05-03 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Lung Neoplasms
Keywords: Awake Thoracic Surgery, Erector Spinae Plane Block
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized between two groups according to loco regional pain management:
  Paravertebral block Erector Spinae Plane Block Allocation to one treatment group or another will be randomized with the aim of create two unbiased groups formed out of the same group of patients. Randomization will be provided by a software.
Who Masked: Participant, Care Provider
Masking Description: Partecipant masking:
  Both blocks are performed on the area between the scapula and the vertebral column, employing the same materials, so that the patient is masked about which block is going to be performed.
  Care providers: once the block has been performed, a different anesthesiologist will take care of the patient during the procedure, eventually providing dose escalation in systemic analgesic drugs (primary end point). Surgeons performing the procedure are unaware of the type of block. Staff nurses managing post operative pain in terms of both recording (Numeric Rating Scale) and soothing (rescue analgesia distribution) are unaware of the type of block (secondary end points).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paravertebral block (PVB) (Active Comparator): Intraoperative pain management
  1. Sedation
     Continuous monitoring of sedation with bispectral index. Sedation is achieved with propofol 1% (target bispectral index: 50-70), plus on-demand remifentanyl (50 mcg/ml in TCI, dose target Cet 2-8 ng/ml).
  2. Paravertebral Block
  Post operative pain management
  * Continuous infusion of Tramadol 200 mg or Ketorolac 60 mg
  * Rescue analgesia with Morphine (0.1 mg/kg) a single time every 24 hours, and/or Tramadol 100 mg up to three times every 24 hours and/ or Ketorolac 30 mg up to three times every 24 hours
  Interventions: Procedure: Paravertebral Block (PVB)
- Erector Spinae Plane Block (ESPB) (Experimental): Intraoperative pain management
  1. Sedation
     Continuous monitoring of sedation with bispectral index. Sedation is achieved with propofol 1% (target bispectral index: 50-70), plus on-demand remifentanyl (50 mcg/ml in TCI, dose target Cet 2-8 ng/ml).
  2. Erector Spinae Plane Block
  Post operative pain management
  * Continuous infusion of Tramadol 200 mg or Ketorolac 60 mg
  * Rescue analgesia with Morphine (0.1 mg/kg) a single time every 24 hours, and/or Tramadol 100 mg up to three times every 24 hours and/ or Ketorolac 30 mg up to three times every 24 hours
  Interventions: Procedure: Erector Spinae Plane Block (ESPB)

INTERVENTIONS:
Procedure: Paravertebral Block (PVB) — PVB consists in the injection of low concentration Ropivacaine (30 ml, 0.3%) in the paravertebral space (defined by the anterior aspect of the ribs, the vertebral body and the parietal pleura. The space is identified under ultrasonographic guidance by a dedicated Anesthesiologist.
  Arms: Paravertebral block (PVB)
Procedure: Erector Spinae Plane Block (ESPB) — ESPB consists in the injection of low concentration Ropivacaine (30 ml, 0.3%), in the anatomical plane between the Erector Spinae muscles and deeper surface of Rhomboid muscle. The space is identified under ecographic guidance, laterally to the spinous process of T5. The diffusion of the anesthetic solution along the space can be echographically appreciated.
  Arms: Erector Spinae Plane Block (ESPB)

SUMMARY:
A randomized prospective trial to test the non-inferiority of Erector Spinae Plane Block (ESPB) in comparison with paravertebral block during non-intubated thoracoscopic lung resection

DETAILED DESCRIPTION:
A prospective randomized trial which aims to evaluate a new technique of peripheral nerve block for pain management, the Erector Spinae Plane Block (ESPB) in patients undergoing minimally invasive lung resection in spontaneous breathing, with intravenous sedation ("non-intubated thoracic surgery"). ESPB will be compared with a largely employed procedure for loco regional pain management: the Paravertebral block (PB). Both procedures are performed under ultrasonographic guidance to allow proper visualization of the target site. Surgery is carried out by means of a minimally invasive approach (Video Assisted thoracic Surgery) with two keyhole incisions on the affected side.

ELIGIBILITY:
Inclusion Criteria:

Wedge Resection of pulmonary nodules performed with a two-portal or three-portal VATS approach.

Peripheral (within 3 cm from the surface of the inflated lung) nodules, less than 2 cm in diameter.

Acceptance of awake VATS with written informed consent

Exclusion Criteria:

Age < 18 years

Patients who are pregnant or lactating

Morbid obesity (BMI > 35 )

Inability to understand and sign the Informed consent

Proven allergy to local anesthetic drugs as required by this protocol

Expected pleural adhesions (previous thoracic trauma, previous pleuro-pulmonary infection, redo surgery on the affected side)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
Dose Escalation of systemic anesthetics during the procedure | 1 hour from the end of the procedure
  Percentage of patients who need sedation escalation

SECONDARY OUTCOMES:
Post operative pain perception | 8, 16, 24 hours from the end of procedure
  Peak pain perception in three time frames (eight hours each) starting from the end of the procedure and covering the first 24 hours after the procedure
Post operative pain management | 8, 16, 24 hours from the end of procedure
  Number of extra doses of rescue analgesia during the first 24 hours after the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Sacro Cuore - Don Calabria Hospital, Negrar, Verona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pompeo E, Mineo D, Rogliani P, Sabato AF, Mineo TC. Feasibility and results of awake thoracoscopic resection of solitary pulmonary nodules. Ann Thorac Surg. 2004 Nov;78(5):1761-8. doi: 10.1016/j.athoracsur.2004.05.083. PMID 15511470
- [Background] Hung MH, Hsu HH, Chan KC, Chen KC, Yie JC, Cheng YJ, Chen JS. Non-intubated thoracoscopic surgery using internal intercostal nerve block, vagal block and targeted sedation. Eur J Cardiothorac Surg. 2014 Oct;46(4):620-5. doi: 10.1093/ejcts/ezu054. Epub 2014 Feb 28. PMID 24585550
- [Background] Liu J, Cui F, Pompeo E, Gonzalez-Rivas D, Chen H, Yin W, Shao W, Li S, Pan H, Shen J, Hamblin L, He J. The impact of non-intubated versus intubated anaesthesia on early outcomes of video-assisted thoracoscopic anatomical resection in non-small-cell lung cancer: a propensity score matching analysis. Eur J Cardiothorac Surg. 2016 Nov;50(5):920-925. doi: 10.1093/ejcts/ezw160. Epub 2016 May 10. PMID 27165771
- [Background] Broseta AM, Errando C, De Andres J, Diaz-Cambronero O, Ortega-Monzo J. Serratus plane block: the regional analgesia technique for thoracoscopy? Anaesthesia. 2015 Nov;70(11):1329-30. doi: 10.1111/anae.13263. No abstract available. PMID 26449303
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Scarfe AJ, Schuhmann-Hingel S, Duncan JK, Ma N, Atukorale YN, Cameron AL. Continuous paravertebral block for post-cardiothoracic surgery analgesia: a systematic review and meta-analysis. Eur J Cardiothorac Surg. 2016 Dec;50(6):1010-1018. doi: 10.1093/ejcts/ezw168. Epub 2016 May 30. PMID 27242357